CLINICAL TRIAL: NCT06862843
Title: Study on Eating Habits and Association with "omic" Profiles in Families with a Subject Affected by a Chronic Immune-mediated Inflammatory Pathology. Observational Multicenter Study.
Acronym: DIETA-MICIREUM
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Paolo Lionetti, Principal Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: DIETA-MICIREUMA
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Juvenile Idiopathic Arthritis (JIA); Crohn Disease (CD); Ulcerative Colitis (UC)
Keywords: JIA; Dietary habits; CD; UC; IBD
MeSH Terms: conditions — Arthritis, Juvenile; Crohn Disease; Colitis, Ulcerative; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples Fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group: Families with at least a member affected with JIA or IBD (UC or CD)
  Interventions: Other: Collecting questionnaires and biological samples
- Control group: Families with all healty components
  Interventions: Other: Collecting questionnaires and biological samples

INTERVENTIONS:
Other: Collecting questionnaires and biological samples — For each family member will be collected a 3-days food diary, a food frequencies questionnaire and a questionnaire assessing the adherence to the mediterranean diet. Additionally, a blood sample for trascriptomic analysis and a fecal sample for gut microbiota analysis will be collected

SUMMARY:
The proposed study is part of a PNRR 2022 project (call "Non-Communicable Chronic Diseases (NCDs) with high impact on healthcare and social assistance systems," currently awaiting funding response) and represents the continuation of an observational clinical study named TRANSMIC, approved by the pediatric ethics committee of the Tuscany region. TRANSMIC was an integral part of a European research project within the joint programming initiative (JPI), under the HDHL-INTIMIC theme: "A Healthy Diet for a Healthy Life," aimed at understanding the cause-effect relationships between diet, gut microbiome, and human health.

Understanding the role of diet in inflammatory bowel diseases (IBD) and exploring its role in autoimmune inflammatory conditions with joint manifestations, such as JIA, provides additional insights into the development, progression, and management of these conditions, opening new horizons for the use of dietary treatments in preventing these inflammatory conditions.

ELIGIBILITY:
Inclusion Criteria:

For families with at least one child/adult affected by IBD/JIA:

* Father and mother with children aged between 0-18 years, in good health.
* At least one adult or one child affected by IBD, or a child affected by JIA, regardless of ongoing therapy and without distinction of disease severity or activity.

For healthy families:

- Father and mother with children aged between 0-18 years, in good health and not affected by chronic inflammatory bowel diseases or chronic autoimmune inflammatory diseases in general.

Exclusion Criteria:

For subjects affected by IBD:

* Monogenic disease
* Children with an ileostomy or who have undergone a colectomy

For subjects affected by JIA:

- No exclusion criteria

For healthy subjects:

- Any chronic inflammatory bowel disease, autoimmune disease, or ongoing infectious diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cases: Families consisting of father, mother, and children aged between 0 and 18 years, in good health, with at least one member (child or adult) affected by IBD (Crohn's disease or ulcerative colitis), and families with a child affected by JIA.
  Controls: Healthy families consisting of father, mother, and children aged between 0 and 18 years, in good health, and not affected by chronic inflammatory bowel diseases or any chronic autoimmune inflammatory diseases.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
3-days food diary, kidmed and medi-lite scores | After two weeks

SECONDARY OUTCOMES:
Percentage of families with microbiota alteration | After 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - AOU Meyer IRCCS, Florence, Italy
  - Università La Sapienza di Roma, Roma, Roma
  - Università di Foggia, Foggia
  - Ospedale Villa Sofia Cervello, Università di Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No